CLINICAL TRIAL: NCT06950450
Title: The Effect of Emotional Freedom Technique (EFT) on Anxiety Experienced Before First Clinical Experience in Nursing Students: A Randomized Controlled Study
Brief Title: EFT and First Clinical Experience Anxiety for Nursing Student
Acronym: EFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Merve Meşedüzü, LECTURER, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-54022451-050.04-184309; MMeseduzu (Other: BezmialemVU)
Record Dates: First submitted 2025-03-03; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: ANXİETY; EFT; CLİNİCAL EXPERİENCE; NURSİNG STUDENT
Keywords: ANXİETY; EFT; NURSİNG STUDENT
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERİMENTAL: EFT GROUP (Experimental): Intervention Group Procedure Steps:
  Pre-Procedure:
  Nursing students in the intervention group will be informed about Emotional Freedom Techniques (EFT), and after explaining the purpose and method of the study, their consent will be obtained using the Volunteer Consent Form.
  They will be asked to complete the Visual Analog Scale (VAS) and State-Trait Anxiety Inventory (STAI) (state-trait version) forms.
  Afterwards, information about EFT will be provided, including how to perform the technique and how to carry out the tapping procedure. After a discussion that is expected to last about 20 minutes, the EFT session will begin. Before the procedure, nursing students will complete the Descriptive Information Form, the State-Trait Anxiety Inventory (STAI-I), and the VAS score forms.
  1. EFT Procedure Sequence: Nursing students who meet the inclusion criteria, including first-year nursing students with no previous clinical experience, will have an initial meeting before their first clini
  Interventions: Behavioral: EMOTİONAL FREE TECHNIQUE
- CONTROL GROUP (No Intervention): Control Group Procedure Steps:
  Control Group - 1st Meeting (Pre-test):
  Nursing students in the control group will be informed about the study, and after explaining the purpose and method of the study, their consent will be obtained using the Volunteer Consent Form.
  The nursing students will be asked to complete the necessary forms, and those who meet the inclusion criteria will be included in the study.
  The nursing students in the control group will complete the Descriptive Information Form, the State-Trait Anxiety Inventory (STAI I-II), and the Visual Analog Scale (VAS) score forms.
  No intervention will be performed for the control group. Instead, the institution's clinical experience procedures will be presented to them.
  Control Group - 2nd Meeting:
  One week after the first meeting and the first clinical experience, the control group nursing students will again complete the State-Trait Anxiety Inventory (STAI I-II) and VAS score forms.
  Control Group - 3rd Meeting:
  Two weeks

INTERVENTIONS:
Behavioral: EMOTİONAL FREE TECHNIQUE — Intervention Group Procedure Steps:
  Pre-Procedure:
  Nursing students in the intervention group will be informed about Emotional Freedom Techniques (EFT), and after explaining the purpose and method of the study, their consent will be obtained using the Volunteer Consent Form.
  They will be asked to complete the Visual Analog Scale (VAS) and State-Trait Anxiety Inventory (STAI) (state-trait version) forms.
  Afterwards, information about EFT will be provided, including how to perform the technique and how to carry out the tapping procedure. After a discussion that is expected to last about 20 minutes, the EFT session will begin. Before the procedure, nursing students will complete the Descriptive Information Form, the State-Trait Anxiety Inventory (STAI-I), and the VAS score forms.
  1. EFT Procedure Sequence: Nursing students who meet the inclusion criteria, including first-year nursing students with no previous clinical experience, will have an initial meeting before their first clinic
  Arms: EXPERİMENTAL: EFT GROUP

SUMMARY:
It was planned as a randomized controlled study to determine the effect of Emotional Freedom Technique (EFT) on Nursing Students' Pre-First Clinical Experience Anxiety.

DETAILED DESCRIPTION:
Clinical experience has been defined by nursing students as one of the most anxiety-inducing components of nursing education. Lack of clinical experience, unfamiliar areas, difficult patients, fear of making mistakes, fear of being evaluated by instructors, and communication issues with hospital staff have been identified by students as situations that cause anxiety during their clinical experiences. Clinical learning experience is a complementary and essential part of nursing education because it enables nursing students to acquire the necessary professional knowledge and skills. It also develops psychomotor skills, which form the foundation for the roles that foster their socialization. This situation can negatively affect the student's clinical performance. Therefore, reducing anxiety and stress levels before the first clinical experience is crucial at every stage of the clinical learning experience . When reviewing studies aimed at reducing nursing students' anxiety before their first clinical experience, methods such as clinical orientation training, pre-clinical simulation, and laboratory training, as well as the use of technology such as artificial intelligence and mobile applications, have been observed.

Gary Craig, an American engineer, developed EFT (Emotional Freedom Techniques) inspired by Roger Callahan's Thought Field Therapy (TFT) . In 1980, Callahan conducted a study on a patient who had a fear of water, causing headaches and nightmares. By tapping on the point below the eyes, which corresponds to the stomach meridian, he discovered that the fear of water was eliminated along with the emotional intensity and fear. He named this approach "Thought Field Therapy" (TFT) . Later, in 1991, Craig conducted research on TFT and, after five years of study, developed a single EFT method that encompasses all conditions .

EFT, an acronym for "Emotional Freedom Techniques," is a psychophysiological intervention that combines somatic stimulation elements using cognitive-behavioral therapy, exposure therapy, and acupuncture points. EFT is an acupressure method designed to improve psychological conditions such as anger, sadness, and anxiety by applying pressure to the meridian points of the organs responsible for these emotions . This method combines traditional psychotherapy with the stimulation of Eastern meridian and acupuncture points, based on the principle of ensuring the smooth flow of energy . EFT is an intervention where a person focuses their physical or psychological awareness on a particular issue while simultaneously tapping on selected acupuncture points, especially on the head and upper torso, with their fingertips . The purpose of this tapping is to create a frequency between the physical body and the energy body, aiming to address the original event that caused the negative emotional state. To achieve full well-being, it is essential to eliminate the energy imbalances caused by the original event that led to the illness .

EFT can be safely used for individuals of all age groups, including children, pregnant women, and the elderly. It can be applied to children for issues like fear, exam stress, nighttime bedwetting, learning difficulties, school anxiety, and eating disorders . In medical conditions, it is used for problems like headaches, physical pain, sleep disorders, constipation, hypertension, respiratory issues, menstrual problems, pregnancy-related nausea, migraines, seizures, and chronic disease symptoms. When using the EFT technique, the Subjective Units of Experience (SUE) scale is used to determine how significant the emotional issue or problem is for the individual. On a scale from -10 to +10, -10 represents the worst possible pain, frustration, fear, stress, sadness, or discomfort (very bad/negative), while +10 represents the highest level of joy, happiness, or feeling great (positive/healing). The tapping used during EFT, also known as Emotional Freedom Technique, is applied to stimulate acupuncture points .

Since EFT is known to reduce anxiety and stress caused by factors such as fear and phobias, it is expected that applying EFT to nursing students about to experience their first clinical experience will reduce their anxiety levels. Based on this hypothesis, this study aims to evaluate the effect of Emotional Freedom Techniques (EFT) on the anxiety levels of nursing students before their first clinical experience through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students in the first year of the BVU SBF Nursing program with a State-Trait Anxiety Inventory (STAI-I, state) score of 20 or higher.

Nursing students with no clinical experience. Nursing students who agree to participate in the study.

Exclusion Criteria:

* tudents enrolled in departments other than the Nursing program. Nursing students in the 2nd, 3rd, or 4th year. Nursing students from different universities.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
EFT AND ANXİETY | 3 months
  H1: Emotional Freedom Technique (EFT) applied to first-year nursing students significantly reduces anxiety levels before clinical practice, as measured by the State-Trait Anxiety Inventory (STAI).
  H2: Emotional Freedom Technique (EFT) applied to first-year nursing students has no significant effect on anxiety levels before clinical practice, as measured by the State-Trait Anxiety Inventory (STAI).
  Title:
  Anxiety Level Before Clinical Practice, Assessed by the State-Trait Anxiety Inventory (STAI)
  Description:
  Anxiety levels will be measured using the State-Trait Anxiety Inventory (STAI), Form Y-1, a widely used 20-item self-report questionnaire designed to assess situational (state) anxiety.
  Participants respond to items based on how they feel "right now, at this moment." Each item is scored on a 4-point Likert scale, resulting in a total score ranging from 20 to 80, where higher scores indicate greater anxiety.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Emotional Free Technical — https://dergipark.org.tr/tr/pub/ybpd/issue/32811/383026